CLINICAL TRIAL: NCT06663579
Title: The Effect of Kangaroo Care Method On The Self-Confıdence and Attachment Levels of Fathers of Preterm Babies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Selmin Kose, Assoc. Prof., Biruni University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Biruni Universitesi
Record Dates: First submitted 2024-10-17; First posted 2024-10-29 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2024-05

CONDITIONS: Attachment Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study group: Fathers who practicing kangaroo care (Experimental): The premature babies treated in the neonatal intensive care unit where the study was conducted practice kangaroo care with their mothers. However, in the intervention conducted by the researcher, the babies practiced kangaroo care with both their mothers and fathers.
  Interventions: Other: Fathers who practicing kangaroo care
- Control group: Fathers who not practicing kangaroo care (No Intervention): The premature babies treated in the neonatal intensive care unit where the study was conducted practice kangaroo care with their mothers. However, in the intervention conducted by the researcher, the babies practiced kangaroo care with both their mothers and fathers.

INTERVENTIONS:
Other: Fathers who practicing kangaroo care — The study group (n=28) It consists of fathers of babies practicing Kangaroo Care with both their mothers and fathers in the neonatal intensive care unit.
  Arms: Study group: Fathers who practicing kangaroo care

SUMMARY:
This study was conducted as a randomized controlled experimental type to evaluate the confidence and attachment levels of fathers in baby care whose babies were treated in the neonatal intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

For Newborns:

* Being a newborn treated in the Istanbul Başakşehir Çam and Sakura Hospital Neonatal Intensive Care Unit
* Gestational age less than 37 weeks
* Postnatal age between 0-28 days
* The baby is considered stable by a neonatologist
* The baby can maintain body temperature during Kangaroo Care
* Safety is ensured if there is an existing umbilical or central catheter

For fathers:

* Agreeing to practice Kangaroo Care
* Having no health condition that would prevent practicing Kangaroo Care
* Being able to maintain sufficient hygiene conditions for Kangaroo Care
* Being literate
* Being able to communicate in Turkish

Exclusion Criteria:

For babies:

* Receiving respiratory support
* Having a chest tube
* Having a congenital anomaly
* Using sedative medication
* Having undergone surgery

For fathers:

* Not wanting to practice Kangaroo Care
* Using substances that cause sedation (drugs, alcohol)
* Having a disease that can be transmitted through skin contact
* Not agreeing to participate in the study
* Not living in the same house as the baby

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2023-11-28 (Actual); Primary Completion 2024-05-28 (Actual); Study Completion 2024-05-28 (Actual)

PRIMARY OUTCOMES:
Paternal-Infant Attachment Scale | This assessment scale will be administered to the father one month following the baby's discharge from the hospital.
  The scale developed to assess father-infant bonding after birth is a 19-item scale. It consists of three subdimensions: 'patience and tolerance,' 'enjoyment in interaction,' and 'love and pride'. Twelve items in the scale are reverse-coded. Higher scores indicate a higher level of bonding. While the original version of the scale consists of 19 items, the Turkish version comprises 18 items. The Cronbach's alpha coefficient of the scale was reported to be 0.81 at 6 months and 0.78 at 12 months.

SECONDARY OUTCOMES:
Karitane Parenting Confidence Scale | This assessment scale will be administered to the father one month following the baby's discharge from the hospital.
  The scale, originally developed by Crncec and colleagues in 2008, was adapted into Turkish by Yılmaz and Oskay in 2021. It is used to assess the self-confidence of parents regarding their parenting abilities and consists of 14 items designed for parents with infants aged 0 to 12 months. The scale includes two sub-dimensions: "Infant Care" and "Parenting Role." Only Item 11 is reverse scored, with the following scoring pattern: 0 = 3; 1 = 2; 2 = 1; 3 = 0. The total score ranges from 0 to 42, with higher scores indicating a more positive outcome and reflecting higher levels of parental self-confidence.

CONTACTS AND LOCATIONS:
Locations (1):
- Biruni University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Due to Hospital policy, the individual participant data can not be shared with anyone except researchers.